CLINICAL TRIAL: NCT03133013
Title: A Study on Realization of Objective Evaluation Method of Depression Using Sleep EEG
Brief Title: Objective Evaluation of Depression Using Sleep EEG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Clete A. Kushida, Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 41103
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with Untreated Depression (Experimental): 32 participants diagnosed with Major Depressive Disorder by a psychiatric specialist of this research according to MINI screening and Diagnostic and Statistical Manual (DSM-5) criteria, and defined as a score of 15 or higher on the clinician-administered Hamilton Rating Scale for Depression, Beck Depression Inventory, and Patient Health Questionnaire for Depression (PHQ-9). The participants will be attached to the SLEEPSCOPE device.
  Interventions: Device: SLEEPSCOPE
- Healthy Participants (Other): 32 healthy participants with absence of mental disorders, including but not limited to depression and sleep disorders, by a psychiatric specialist according to MINI screening and Diagnostic and Statistical Manual (DSM-5) criteria, and negative Hamilton Rating Scale for Depression, Beck Depression Inventory, and Patient Health Questionnaire for Depression (PHQ-9). The participants will be attached to the SLEEPSCOPE device.
  Interventions: Device: SLEEPSCOPE

INTERVENTIONS:
Device: SLEEPSCOPE — Brainwave measurement device which is connected to the participant by an electrode attached to the forehead and another electrode behind one ear

SUMMARY:
The purpose of this study is to test the ability of a brainwave measurement device (SLEEPSCOPE) in identifying and assisting in the diagnosis of depression. The brainwave data from individuals with untreated depression and healthy participants will be collected and analyzed. The ability to obtain brainwave data from individuals in their homes while they're sleeping would represent a significant advance in depression research.

DETAILED DESCRIPTION:
The purpose of study is to collect and analyze human sleeping brainwave data, to better understand depression in humans.

First visit:

* Informed consent procedures, including explanation of research background, purpose, details of implementation, and study benefits and risks
* Interview with questionnaires (MINI International Psychiatric Interview, Hamilton Rating Scale for Depression, Beck Depression Inventory, Patient Health Questionnaire for Depression [PHQ-9]), physical examination.
* Urine drug sample for screening of controlled substances.
* Inform participants that those qualifying will be informed whether or not to proceed with second visit

Second visit:

* Explanation of EEG measurement (placement of two electrodes, one on the forehead and one behind the ear)
* Sleep diary provided for participant to complete at home for each night until third visit
* Distribution of EEG devices for home use
* EEG measurement conducted at participant's residence for three nights of stable sleep-wake cycles

Third visit:

- Collect EEG devices and check completeness of downloaded data

ELIGIBILITY:
Inclusion Criteria:

Individuals with Untreated Depression:

- 16 men and 16 women aged from 30 to 59 years, with an approximate ethnic balance of 10 Asian, 3 White and 3 other ethnicity for each gender, whom are diagnosed with Major Depressive Disorder by a psychiatric specialist of this research according to MINI screening and DSM-5 criteria, and defined as a score of 15 or higher on the clinician-administered Hamilton Rating Scale for Depression, Beck Depression Inventory, and Patient Health Questionnaire for Depression (PHQ-9).

Healthy Participants:

- 16 men and 16 women age-, ethnic-, and gender-matched healthy participants to the cohort with untreated depression, with absence of mental disorders, including but not limited to depression and sleep disorders, by a psychiatric specialist according to MINI screening and DSM-5 criteria, and negative Hamilton Rating Scale for Depression, Beck Depression Inventory, and Patient Health Questionnaire for Depression (PHQ-9).

Exclusion Criteria:

Participants corresponding to any of the following conditions are considered ineligible for the trial.

* Diagnosed with epilepsy or other organic brain disorder.
* Medical conditions resulting in depressive symptoms such as hypothyroidism, Cushing's disease, systemic lupus erythematosus; neurological conditions resulting in depressive symptoms such as Parkinson's disease, Huntington's disease, multiple sclerosis
* Patients with suspected sleep apnea, based on symptoms and a BMI of 30 or greater
* Prescribed interferon regularly with stimulants, opioid drugs (Ritalin, Opioid, etc.) and steroids
* Repetitive thoughts of death, current thoughts about suicide, suicide attempts, or a suicide plan
* Tested positive to controlled substance use by a urine drug screening before commencement of testing
* Current or past drug or alcohol dependence
* Shift work or rotating work schedule
* Nursing, pregnant or planning to become pregnant
* Participating in other clinical trials

Ages: 30 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Assist in the diagnosis of depression | 1 month
  The SLEEPSCOPE data will be analyzed to determine if it can help to identify individuals with depression

CONTACTS AND LOCATIONS:
Overall Officials: Clete A Kushida, M.D., Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Sleep Medicine Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No